CLINICAL TRIAL: NCT03944148
Title: Thoracic Point of Care Ultrasound on Initial Management of Upper Gastrointestinal Bleeding
Brief Title: Thoracic Ultrasound on Upper Gastrointestinal Bleeding (ECOBLEDSTUDY)
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Dr. med. Hector Eloy Tamez Perez, Clinical Professor, Hospital Universitario Dr. Jose E. Gonzalez
Other Study IDs: G19-00001
Record Dates: First submitted 2019-04-16; First posted 2019-05-09 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Upper Gastrointestinal Bleeding
Keywords: Upper Gastrointestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Upper Gastrointestinal bleeding (UGIB) is a medical emergency and the most common cause of hospitalization associated with digestive disease. Proper initial resuscitation is the first step in the management of UGIB patients. Today, modern pulmonary ultrasound is used in different clinical settings, such as intensive care, emergency medicine and/or traumatology. In the last years, the use of this has been standardized both in internal medicine and in pulmonary medicine. The primary objective is to describe the findings of pulmonary ultrasound and its relationship with severity in patients with UGIB. The investigators will include all patients with UGIB. A pulmonary and vena cava ultrasound will be performed on admission to the emergency room, 10 minutes prior to endoscopy and 24 hours after having performed the endoscopy.

The use of thoracic point-of-care ultrasound (TPOCUS) has been standardized in both internal and pulmonary medicine. There is a concern about the role of TPOCUS useful as a severity prognostic tool in patients with UGIB.

The team proposes that TPOCUS is a severity prognostic tool in UGIB patients.

Main Outcome: To describe the findings of TPOCUS in patients with variceal and non-variceal UGIB.

Secondary Objectives:

1. Correlate the presence of B-type lines on TPOCUS with mean arterial pressure in UGIB patients.
2. Correlate the inferior vena cava diameter with the Model for End-stage Liver Disease scale in UGIB patients.
3. Correlate the inferior vena cava diameter with the 48 hours post-admission mortality of UGIB patients.

Authors design a prospective, longitudinal, descriptive study to identify the findings of TPOCUS in patients with variceal and non-variceal UGIB. Patients will be included in the study since May 15th through October 30th 2019, admitted to the University Hospital, "Dr. José E. González", Universidad Autónoma de Nuevo León.

DETAILED DESCRIPTION:
Inclusion criteria:

1. Patients with a diagnosis of UGIB documented by endoscopy.
2. Any gender.
3. Over 18 years old.

Exclusion criteria:

1. Patients with UGIB previously treated in other hospitals.
2. Patients under 18 years of age.
3. Patients with suspected UGIB who did not undergo endoscopy.
4. Pregnant.
5. Patients with chronic obstructive pulmonary disease.
6. Patients with interstitial lung disease.
7. Patients with pleural effusion at the time of admission to the emergency room.
8. Refusal to participate in the protocol.

Method The investigators will study all patients who come to the emergency room of the hospital due to suspicion of UGIB (melena, hematemesis, vomiting in coffee grounds and hematochezia with hemodynamic instability). These patients will undergo a pulmonary and vena cava ultrasound.

Patients with suspected UGIB who are candidates for upper endoscopy during their hospital stay will undergo a second pulmonary and vena cava ultrasound ten minutes prior to upper endoscopy.

The investigators will include in the research study patients with UGIB documented by upper endoscopy. The investigators will perform a third pulmonary and vena cava ultrasound 24 hours after the endoscopic procedure.

The investigators will exclude patients with suspected UGIB but who are not candidates for endoscopy.

The technique used is a bilateral intercostal thoracic point-of-care ultrasound (TPOCUS) with the patient in supine decubitus with the head at 30 degrees. Each hemithorax will be divided into 4 areas: anterior and lateral, superior and inferior. The anterior area will be delineated between the clavicle and the diaphragm and between the parasternal line to the anterior axillary line. The lateral area will be delineated between the axilla and the diaphragm and between the anterior to the posterior axillary line. The superior area will be delineated from the 1st to the 3rd intercostal space and the lower area from the 4th to the 6th intercostal space. A total of 8 areas of the chest will be visualized during normal breathing.

The TPOCUS findings to report are:

B-type lines: Those lines are hydro-aerial artifacts presenting as comet tail images, begin in the pleural line, are hyper-echoic, well defined, disseminated towards the end of the screen, delete A-type lines, and move with the pleural slip when this it is present. The lines separated from each other around 7 mm correspond to interstitial edema, while those that distance 3 mm indicate the presence of alveolar edema. The presence of more than 3 B-type lines indicates the presence of an alveolar-interstitial syndrome.

The inferior cava vein evaluation will be performed by measuring the diameter and percentage of collapse of this vein. It will be performed in the subxiphoid window with the identification of the four cardiac chambers, then a 90º turn of the transducer will made in the cephalad direction, which will show the right atrium, the union of the inferior vena cava and the liver above it. The diameter measurement will be beyond the point of confluence of the hepatic veins, usually found approximately 2 cm from the union of the inferior vena cava and the right atrium. Based on the diameter and collapse percentage measurement of the inferior vena cava on spontaneous breathing, a volume status will be defined as lack of volume if the diameter is <2 cm and the collapse percentage is >50%; however, a diameter >2 cm and a collapse percentage <50% will be classified as hypervolemic state.

ELIGIBILITY:
Inclusion Criteria:

* Age, more than 17 years old.
* Patients diagnosed with UGIB.
* Any etiology of the UGIB.

Exclusion Criteria:

* Patients with UGIB previously treated in other hospitals.
* Patients with UGIB with Blatchford scale less than 2 points.
* Pregnant women.
* Refusal to participate in the protocol.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with variceal and non-variceal UGIB, who arrive to the emergency department of the University Hospital, "Dr. José E. González" Universidad Autónoma de Nuevo León.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
B-type lines on thoracic point-of-care ultrasound in patients with UGIB. | 48 hours
  The number of B-type lines measured by thoracic point-of-care ultrasound in patients with variceal and non-variceal UGIB at 48 hours.
Diameter of inferior vena cava on thoracic point-of-care ultrasound in patients with UGIB. | 48 hours
  The diameter in centimeters of inferior vena cava measured by thoracic point-of-care ultrasound in patients with variceal and non-variceal UGIB at 48 hours.

SECONDARY OUTCOMES:
B-type lines and mean arterial pressure on UGIB patients | 48 hours
  To correlate the presence of B-type lines on thoracic point-of-care ultrasound with mean arterial pressure in UGIB patients.
Inferior vena cava diameter and Model for End-stage Liver Disease on UGIB patients | 48 hours
  To correlate the inferior vena cava diameter with the Model for End-stage Liver Disease scale in UGIB patients.
Inferior vena cava diameter and 48 hours mortality in UGIB patients. | 48 hours
  To correlate the inferior vena cava diameter with the 48 hours post-admission mortality rate in UGIB patients.

CONTACTS AND LOCATIONS:
Overall Officials: Hector Ibarra Sifuentes, M.D., Principal Investigator — Universidad Autonoma de Nuevo Leon
Locations (1):
- Hospital Universitario Dr. Jose E. Gonzalez, Universidad Autónoma de Nuevo León, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Yes
If need information will be available upon email contact request.
Supporting Information: Study Protocol
Time Frame: 1 year
Access Criteria: email contact request for academic purposes.